CLINICAL TRIAL: NCT04431401
Title: Repetitive Transcranial Magnetic Stimulation in the Treatment of Primary Progressive Aphasia: A Randomized Controlled Trial
Brief Title: rTMS Treatment of Primary Progressive Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPA-rTMS
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-03

CONDITIONS: Primary Progressive Aphasia; Repetitive Transcranical Magnetic Stimulation
MeSH Terms: conditions — Aphasia, Primary Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS treatment group (Experimental): The participants will be divided into the rTMS treatment group and the sham treatment group by means of randomized methods.The protocol of the treatment is to use rTMS with high frequency 10/20Hz 120%RMT 20 times for one month. The device is Magtism rTMS made in London, UK
  Interventions: Device: Magstim rTMS
- sham treatment group (Sham Comparator): The control group is to receive sham treatment. The device is the same as the one used in the real treatment group.
  Interventions: Device: Magstim rTMS

INTERVENTIONS:
Device: Magstim rTMS — The device is made in London,UK

SUMMARY:
Primary Progressive Aphasia (PPA) is a neurodegenerative disease in which language function is gradually and progressively impaired. Patients will eventually be disabled in communication and have cognition deficits, which put a heavy burden not only on their families but also on the whole society. However, no effective treatment for PPA has been explored so far. The current clinical randomized trial is to study the safety and efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) for the treatment of PPA. Also, multi-modality of neuroimaging techniques, such as functional MRI and PET will be used to investigate brain network changing in this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PPA

Exclusion Criteria:

* Scored below 15 on the mini-mental state exam (MMSE)
* history of seizures or unexplained loss of consciousness
* pregnancy
* surgical breach of the skull
* MRI contraindication

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Boston naming test evaluation | 1 day before the treatment
  Assessment of the language production. Scores range from 0 to 30. Higher scores means better outcome.
Boston naming test evaluation | 1 month, 3 months and 6 months after the treatment
  Assessment of the language production. Scores range from 0 to 30. Higher scores means better outcome.
Western Aphasia Battery (WAB) Speech fluency | 1 day before the treatment
  Assessment of the language production. Scores range from 0 to 20. Higher scores means better outcome.
Western Aphasia Battery (WAB) Speech fluency | 1 month, 3 months and 6 months after the treatment
  Assessment of the language production. Scores range from 0 to 20. Higher scores means better outcome.
Western Aphasia Battery (WAB) Repetition | 1 day before the treatment
  Assessment of the repetition ability. Scores range from 0 to 100. Higher scores means better outcome.
Western Aphasia Battery (WAB) Repetition | 1 month, 3 months and 6 months after the treatment
  Assessment of the repetition ability. Scores range from 0 to 100. Higher scores means better outcome.
Western Aphasia Battery (WAB) Word recognition | 1 day before the treatment
  Assessment of the reading. Scores range from 0 to 60. Higher scores means better outcome.
Western Aphasia Battery (WAB) Word recognition | 1 month, 3 months and 6 months after the treatment
  Assessment of the reading. Scores range from 0 to 60. Higher scores means better outcome.
Syntax comprehension part of Bilingual aphasia test (Standard Modern Chinese Version) | 1 day before the treatment
  Assessment of the grammar ability. Scores range from 0 to 50. Higher scores means better outcome.
Syntax comprehension part of Bilingual aphasia test (Standard Modern Chinese Version) | 1 month, 3 months and 6 months after the treatment
  Assessment of the grammar ability. Scores range from 0 to 50. Higher scores means better outcome.

SECONDARY OUTCOMES:
functional connectivity map (FC map) | 1 day before the treatment
  Functional Connectivity was examined using a seed-based voxel-wise correlation approach. The language related brain areas, such as Broca Area and Wernicke Area, were defined as the regions of interest (ROI). Pearson's correlation analysis between the time course of the ROI and that of every voxel in the whole brain was computed for a map of correlation coefficients, which were Fisher's z-transformed and called as z-FC maps. This outcome measurement, the z-FC map, is not numeric data. Z-FC map is a radiographic imaging measurement.
functional connectivity map (FC map) | 1 month, 3 months and 6 months after the treatment
  Functional Connectivity was examined using a seed-based voxel-wise correlation approach. The language related brain areas, such as Broca Area and Wernicke Area, were defined as the regions of interest (ROI). Pearson's correlation analysis between the time course of the ROI and that of every voxel in the whole brain was computed for a map of correlation coefficients, which were Fisher's z-transformed and called as z-FC maps. This outcome measurement, the z-FC map, is not numeric data. Z-FC map is a radiographic imaging measurement.
Standardized Uptake Value (SUV) | 1 day before the treatment
  PET parameter to evaluate brain metabolism
Standardized Uptake Value (SUV) | 1 month, 3 months and 6 months after the treatment
  PET parameter to evaluate brain metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Huang Y, Tan Y, Hao H, Li J, Liu C, Hu Y, Wu Y, Ding Q, Zhou Y, Li Y, Guan Y. Treatment of primary progressive aphasia by repetitive transcranial magnetic stimulation: a randomized, double-blind, placebo-controlled study. J Neural Transm (Vienna). 2023 Feb;130(2):111-123. doi: 10.1007/s00702-023-02594-w. Epub 2023 Jan 20. PMID 36662282